CLINICAL TRIAL: NCT00836550
Title: An RCT to Evaluate the Effectiveness of an Emergency Department Based Multimedia HIV Testing Model in Adolescents
Brief Title: Video-based Counseling & Rapid HIV Testing for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Bronx Healthcare Network (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Yvette Calderon/ Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2005-456-001; HD054315-02
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: HIV; HIV Infections
Keywords: HIV; HIV knowledge measure; Teen HIV testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): The participants spoke with a live counselor prior to answering the knowledge measure
  Interventions: Behavioral: in-person HIV pre-test counseling
- Video (Experimental)
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Video — The participants saw a 6 minute video
  Arms: Video
Behavioral: in-person HIV pre-test counseling
  Arms: Control

SUMMARY:
This study evaluated the educational effectiveness of a youth-friendly pre-test video (derived from a previous qualitative study) and compared it with in-person HIV pre-test counseling. A convenience sample of 200 medically stable individuals between the ages of 15 and 21 presenting to an urban ED were recruited to participate in this study and randomized into 2 groups. Individuals were eligible if they were English-speaking, sexually active and able to consent. All participants completed a sexual risk factor and demographic survey. Group 1 completed a validated pre-test knowledge measure, viewed the HIV education video then completed a post-test knowledge measure. Group 2 completed the same knowledge measures, but received pre-test HIV counseling from a trained public health advocate. HIV testing was optional

ELIGIBILITY:
Inclusion Criteria:

* 15-21 year old
* sexually active
* English-Speaking

Exclusion Criteria:

* medically unstable

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Knowledge of HIV | 2 months

SECONDARY OUTCOMES:
Consent to HIV testing | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD MS, Principal Investigator — Jacobi Medical Center/ Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States